CLINICAL TRIAL: NCT05192434
Title: Efficacy of a Trauma Intervention for Affect Regulation, Adherence, and Substance Use to Optimize PrEP for Women Who Inject Drugs
Brief Title: Trauma Intervention to Optimize PrEP Among Women Who Inject Drugs
Acronym: TIARAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alexis Roth, Associate Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2105008584; R01DA054543 (NIH)
Record Dates: First submitted 2022-01-05; First posted 2022-01-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections; Opioid Use; Trauma, Psychological
Keywords: PrEP; Preexposure Prophylaxis; WWID; Women who inject drugs
MeSH Terms: conditions — HIV Infections; Psychological Trauma

STUDY DESIGN:
Intervention Model Description: Our concurrent nested mixed methods RCT will test the efficacy of addressing trauma as a potent trigger of substance use and psychological comorbidity through Expressive Writing (EW) among WWID receiving Contingency Management (CM). We will enroll 240 WWID who initiate PrEP. After a run-in period, participants will be randomized to either: 1) EW+CM (n=120); or 2) Neutral Writing+CM (n=120).
Who Masked: Investigator
Masking Description: Study personnel who administer survey assessments will be blinded to study participants' assignment to the expressive writing group (treatment) or the neutral writing group (control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive Writing + Contingency Management (Experimental): A total of 120 WWID will be randomly assigned to the EW+CM (expressive writing + contingency management) intervention arm. To begin each session, participants will complete a brief battery of psychological measures. Then, in a private setting, they will be asked to write for 20 minutes about a major trauma that occurred three or more months in the past. WWID who prefer not to write (e.g., have lower literacy) will be provided the opportunity to talk aloud about the traumatic experience while being audio recorded, which yields comparable effects to writing. Next, women will respond to a prompt that encourages cognitive processing of the trauma for ten additional minutes. To complete the session, participants will answer the same brief battery of psychological measures for the purposes of identifying acute distress. Those exhibiting clinically elevated distress symptoms will engage in a brief de-escalation and evaluation session with study staff who will be trained.
  Interventions: Behavioral: Expressive Writing; Behavioral: Contingency Management
- Neutral Writing + Contingency Management (Placebo Comparator): A total of 120 WWID will be randomly assigned to the attention-control arm which includes neutral writing + CM. Women in this group will complete the same pre/post psychological measures as the intervention group for the purposes of time matching. During the writing session, they will be asked to describe their schedule from the preceding day as if they were reporting facts, without discussing personal thoughts and feelings (e.g., describe what you did from the time you got up until the time you went to bed). Those with lower literacy can opt to talk aloud while being audio recorded. This is the same attention-control used our previous work which balances contact time and study incentives.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Expressive Writing — Expressive writing (EW) is a safe, acceptable, and effective intervention for improving psychological adjustment. Via brief directed writing sessions, EW facilitates disclosure of traumatic events. At a basic level, emotional expression and disclosure are important because they reduce the need to unconsciously direct psychological energy towards suppressing emotions from traumatic events.
  Arms: Expressive Writing + Contingency Management
Behavioral: Contingency Management — Contingency management (CM) is a proven strategy to reduce drug use and HIV risk behavior. Also known as a conditional cash transfer, CM reinforces positive behavior with tangible rewards. In the context of substance use treatment, monetary incentives are typically used to reinforce drug-negative urine specimens.

SUMMARY:
The goal of this randomized controlled trial is to test the effectiveness of "TIARAS," a trauma intervention designed to reduce HIV acquisition risk among women who inject drugs (WWID). To be eligible for this study, participants must have been prescribed pre-exposure prophylaxis (PrEP), a medication taken to prevent HIV, at Prevention Point Philadelphia, a large harm reduction agency located in Philadelphia (PA, USA), or Courage Medicine, a nonprofit health services clinic located in Philadelphia (PA, USA).

Enrollment in this study lasts for 12-months so that we can see if TIARAS reduces HIV risk immediately after the intervention ends and whether these effects last over time. During the first 3 months, participants engage in contingency management (CM), an evidenced-based intervention to reduce drug use and HIV risk. We will use CM to encourage engagement in PrEP care as well as stimulant/opioid abstinence. Also during the first 3-months, participants are randomly assigned to complete expressive writing exercises to address a previously undisclosed trauma or neutral writing exercises. Half of the participants will be assigned to the trauma writing group and the other half will be assigned to the neutral writing group.

To understand the impact of TIARAS on HIV risk, we will collect and analyze data from surveys, interviews, and biological specimen during the 12-month study period. Our main questions are:

* Does participation in TIARAS reduce HIV risk among WWID?
* If observed, how long do beneficial effects last?
* How and why do WWID experience benefits from TIARAS?

DETAILED DESCRIPTION:
In the United States, recent outbreaks coast-to-coast forewarn of a possible resurgence of HIV, especially among women who inject drugs (WWID), particularly if access, uptake, and adherence to effective harm reduction tools remain sub-optimal. Pre-exposure prophylaxis (PrEP) is a user-driven method that safely and effectively prevents HIV. While we have shown that cisgender WWID consider PrEP beneficial and are willing to accept a prescription, consistent with the well-known SAVA syndemic framework, social stigma, economic insecurity, traumatic experiences (or the threat of violence), and drug use greatly undermined their agency to prioritize and adhere to PrEP. This trauma-informed randomized control trial (RCT) will address the urgent need for HIV prevention interventions, informed by the SAVA framework, that produce durable reductions in HIV risk among WWID. We will integrate contingency management (CM), a proven strategy to reduce drug use and HIV risk, and expressive writing (EW), a safe and effective approach for addressing trauma symptoms, in order to test whether EW delivered during CM (EW+CM) produces durable reductions in HIV acquisition risk compared to an attention-control condition. We will leverage our partnership with Prevention Point Philadelphia (PPP), the largest syringe exchange in the mid-Atlantic, and Courage Medicine to recruit 240 WWID who will (re)initiate PrEP at PPP or Courage Medicine. Once enrolled they will immediately begin a 3-month CM period that provides incentives for directly observed daily oral PrEP doses or confirmed injectable PrEP doses, stimulant/opioid abstinence (measured thrice weekly through urine screening), and completion of four writing sessions. After a run-in period, WWID will be randomized to either EW+CM (n=120) or Neutral Writing+CM (n=120). Follow-up assessments will occur at 3-, 6-, and 12-months post-randomization and will include objective measures of PrEP adherence over time. A subset of WWID from both arms will complete qualitative interviews at 3- and 12-months. All study activities and daily PrEP dispensing will occur at PPP. The specific aims are to: (1) Determine the efficacy of EW+CM for improving the proportion of participants achieving reductions in HIV acquisition risk (operationalized as the proportion of WWID reporting syringe sharing or condomless sex during objectively measured periods of PrEP non-adherence) at 12 months. (2) Examine key secondary outcomes such as greater PrEP persistence, reductions in substance use, PTSD symptoms, and depression, as well as entry into drug treatment over 12 months. (3) Evaluate the pathways through which the intervention operates using qualitative interviews, mediation analysis (e.g., emotional expression and processing in EW essays), and moderation analysis (e.g., more pronounced among those with higher PTSD severity at baseline). This RCT could have an exceptional impact by yielding one of the first evidence-based interventions to address HIV acquisition risk in the era of PrEP among WWID.

ELIGIBILITY:
Inclusion Criteria:

a) HIV-negative cisgender female, b) age ≥ 18 years, c) speaks/reads English d) reporting past 6 months day non-prescription injection drug use and any of the following: NEW PrEP PATIENT: prescribed daily oral or injectable PrEP at Prevention Point Philadelphia or Courage Medicine within 30 days. For injectable PrEP, they will be considered new if they have received a prescription but are within two weeks of receiving their first injection. or NON-ADHERENT DAILY ORAL PrEP PATIENT: initiated PrEP at Prevention Point Philadelphia or Courage Medicine 30 or more days ago who reports any non-adherence or reports consistent adherence but has PrEP-related drug levels indicating non-adherence (verified with urine-based tenofovir testing) or NON-ADHERENT INJECTABLE PrEP PATIENT: initiated injectable PrEP at Prevention Point Philadelphia or Courage Medicine but is 8 or more days late to receive their next injection (verified in participant's electronic medical record)

Exclusion Criteria:

a) Unable to provide informed consent; b); unwilling or unable to return to the SSP daily for the next 90 days; c) unwilling to provide specimen for PrEP-related clinical monitoring and adherence monitoring; d) pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender females eligible
Enrollment: 219 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HIV Acquisition Risk | Participant duration (1 year)
  Our primary outcome will be a composite of two measures: self-reported behavioral HIV risk (syringe sharing or condomless sex) and objectively measured adherence to PrEP. To assess PrEP adherence in women initiating daily oral Tenofovir-based (TFV) PrEP products, we will collect scalp hair at baseline, 3, 6, and 12 months. Specimens will be tested using liquid chromatography/tandem mass spectrometry to quantify TFV concentrations levels. In primary analysis, and TFV level >/= 0.025.ng, consistent with >/= 6 doses per week, will be considered adherent. To assess PrEP adherence in women initiating cabotegravir PrEP products, we will extract the dates of LAI-CAB injections from participants' electronic medical records and will determine whether each follow-up LAI-CAB injection occurred within recommended dosing windows according to Apretude prescribing information (+/- 7 days). In primary analysis, any injection occurring within the recommended dosing window will be considered adherent.

SECONDARY OUTCOMES:
Reductions in Drug Use | Participation duration (1 year)
  At each study visit, participants will complete The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST), which assesses lifetime and recent (past 90 day) drug use. We will describe recent substance use and determine whether there are clinically meaningful decreases in illicit stimulant and/or opioid use over time.
Drug Abstinence | Participation duration (1 year)
  Participants will provide urine samples for oon-site toxicology screening of methamphetamine, cocaine, and opioid metabolites. Reactive urine toxicology results are indicative of stimulant/opioid use within the past 72 hours. Results of urine drug screens will be extracted from electronic medical records.
Referrals for Drug Treatment | Participation duration (1 year)
  Participant requests for a referral for drug treatment will be captured during study visits and logged into the study database. To calculate the number of referrals, we will extract data from the study database.
Depression | Participation duration (1 year)
  We will use the Beck Depression Inventory (BDI). This validated 21 item scale has a score range of 0 to 63. A cutoff score of 19 will be used to classify moderate/severe depressive symptoms.
PTSD Symptoms | Participation duration (1 year)
  We will use the PTSD checklist from DSM 5 (PCL-5). This is a 20 item validated scale with a score range 0 to 80. This generates 5 sub-scales symptom scores, which will be assessed for particular patterns of symptomology. A total cutoff score ≥ 33 will be used to classify moderate/severe PTSD.
Cost effectiveness | Participation duration (1 year)
  Cost effectiveness will be estimated using a micro-costing approach. Cost offsets will be collected using the Non-Study Medical and Other Services (NMOS) assessment tool along with the Patient Reported Outcomes Measurement Information System (PROMIS PROPr) assessment tool to determine QUALYs. Cost data collection and analysis will be informed by the Drug Abuse Treatment Cost Analysis Program (DATCAP), a standardized costing tool used in hundreds of clinical trials over the past 3 decades.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis M Roth, PhD, MPH, Principal Investigator — Drexel University
Locations (1):
- Prevention Point Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plotzker RE, Metzger DS, Holmes WC. Childhood sexual and physical abuse histories, PTSD, depression, and HIV risk outcomes in women injection drug users: a potential mediating pathway. Am J Addict. 2007 Nov-Dec;16(6):431-8. doi: 10.1080/10550490701643161. PMID 18058406
- [Background] Prendergast M, Podus D, Finney J, Greenwell L, Roll J. Contingency management for treatment of substance use disorders: a meta-analysis. Addiction. 2006 Nov;101(11):1546-60. doi: 10.1111/j.1360-0443.2006.01581.x. PMID 17034434
- [Background] Haug NA, Sorensen JL. Contingency management interventions for HIV-related behaviors. Curr HIV/AIDS Rep. 2006 Nov;3(4):154-9. doi: 10.1007/s11904-006-0010-5. PMID 17032574
- [Background] Rosen MI, Dieckhaus K, McMahon TJ, Valdes B, Petry NM, Cramer J, Rounsaville B. Improved adherence with contingency management. AIDS Patient Care STDS. 2007 Jan;21(1):30-40. doi: 10.1089/apc.2006.0028. PMID 17263651
- [Background] Carrico AW, Nation A, Gomez W, Sundberg J, Dilworth SE, Johnson MO, Moskowitz JT, Rose CD. Pilot trial of an expressive writing intervention with HIV-positive methamphetamine-using men who have sex with men. Psychol Addict Behav. 2015 Jun;29(2):277-82. doi: 10.1037/adb0000031. Epub 2014 Dec 1. PMID 25437153
- [Background] Baikie KA, Wilhelm K, Johnson B, Boskovic M, Wedgwood L, Finch A, Huon G. Expressive writing for high-risk drug dependent patients in a primary care clinic: a pilot study. Harm Reduct J. 2006 Nov 19;3:34. doi: 10.1186/1477-7517-3-34. PMID 17112389
- [Background] Meshberg-Cohen S, Svikis D, McMahon TJ. Expressive writing as a therapeutic process for drug-dependent women. Subst Abus. 2014;35(1):80-8. doi: 10.1080/08897077.2013.805181. PMID 24588298
- [Background] Koopman C, Ismailji T, Holmes D, Classen CC, Palesh O, Wales T. The effects of expressive writing on pain, depression and posttraumatic stress disorder symptoms in survivors of intimate partner violence. J Health Psychol. 2005 Mar;10(2):211-21. doi: 10.1177/1359105305049769. PMID 15723891
- [Background] Ironson G, Bira L, Hylton E. Positive and negative emotional expression measured from a single written essay about trauma predicts survival 17 years later in people living with HIV. J Psychosom Res. 2020 Sep;136:110166. doi: 10.1016/j.jpsychores.2020.110166. Epub 2020 Jun 9. PMID 32559504
- [Background] O'Cleirigh C, Ironson G, Antoni M, Fletcher MA, McGuffey L, Balbin E, Schneiderman N, Solomon G. Emotional expression and depth processing of trauma and their relation to long-term survival in patients with HIV/AIDS. J Psychosom Res. 2003 Mar;54(3):225-35. doi: 10.1016/s0022-3999(02)00524-x. PMID 12614832
- [Background] Ironson G, O'Cleirigh C, Leserman J, Stuetzle R, Fordiani J, Fletcher M, Schneiderman N. Gender-specific effects of an augmented written emotional disclosure intervention on posttraumatic, depressive, and HIV-disease-related outcomes: a randomized, controlled trial. J Consult Clin Psychol. 2013 Apr;81(2):284-98. doi: 10.1037/a0030814. Epub 2012 Dec 17. PMID 23244367
- [Result] Roth AM, Bartholomew TS, Ward KM, Groves A, Mazzella S, Bellamy S, Amico KR, Carrico AW, Ironson G, Krakower D. Preferential Initiation of Long-Acting Injectable Versus Oral HIV Pre-Exposure Prophylaxis Among Women Who Inject Drugs. Clin Infect Dis. 2025 Mar 17;80(3):621-625. doi: 10.1093/cid/ciae450. PMID 39347705
- [Derived] Ward KM, Carrico AW, Vader D, Moore RH, Amico KR, Groves AK, Bellamy SL, Sherman SG, Krakower D, Mazzella S, Roth AM. Implementation of contingency management with women engaging in polysubstance use. Addict Sci Clin Pract. 2025 Aug 8;20(1):63. doi: 10.1186/s13722-025-00590-x. PMID 40781335